CLINICAL TRIAL: NCT01762774
Title: A Single-centre, Randomised, Double-blind, Placebo-controlled, Escalating Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Doses of GSK2256294 in Healthy Volunteers, and Single and Repeat Doses of GSK2256294 in Adult Male Moderately Obese Smokers
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Doses of GSK2256294 in Healthy Volunteers, and Single and Repeat Doses of GSK2256294 in Adult Male Moderately Obese Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 114068
Record Dates: First submitted 2012-12-13; First posted 2013-01-08 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; forearm blood flow; soluble Epoxide Hydrolase inhibitor
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — N-((4-cyano-2-(trifluoromethyl)phenyl)methyl)-3-((4-methyl-6-(methylamino)-1,3,5-triazin-2-yl)amino)cyclohexanecarboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): Healthy male subjects in this cohort will take part in 4 treatment periods with one of the following treatments in each period. Subjects will receive single dose of all four treatments (one per period) in a random order. Treatment A = 2 mg GSK2256294 capsules, Treatment B = 6 mg GSK2256294 capsules, Treatment C = 18 mg GSK2256294 capsules, Treatment P = Matched Placebo capsules.
  Interventions: Drug: GSK2256294; Drug: Placebo
- Cohort 2 (Experimental): Obese adult male smoker subjects in this cohort will take part in 4 treatment periods with one of the following treatments in each period. Subjects will receive single dose of all four treatments (one per period) in a random order. Treatment A = 15 mg GSK2256294 capsules, Treatment B = 40 mg GSK2256294 capsules, Treatment C = 100 mg GSK2256294 capsules, Treatment P = Matched Placebo capsules.
  Interventions: Drug: GSK2256294; Drug: Placebo
- Cohort 3 (Experimental): Obese adult male smoker subjects in Cohort 3 will receive single or twice daily dose of GSK2256294 or placebo for 14 days. Dose selection for Cohort 3 will be based on the safety, PK profile and enzyme inhibition obtained in cohorts 1 and 2.
  Interventions: Drug: GSK2256294; Drug: Placebo
- Cohort 4 (Experimental): Obese adult male smoker subjects in Cohort 4 will receive single or twice daily dose of GSK2256294 or placebo for 14 days. Dose selection for Cohort 4 will be based on the safety, PK profile and enzyme inhibition obtained in cohorts 1 and 2 as well as safety and PK profile obtained in cohort 3.
  Interventions: Drug: GSK2256294; Drug: Placebo

INTERVENTIONS:
Drug: GSK2256294 — GSK2256294 capsules will be administered as once daily as single dose 2 mg, 6 mg, 15 mg in Cohort 1 and 15 mg, 40 mg, 100 mg in Cohort 2. GSK2256294 capsules will be administered once or twice daily (cohorts 3 and 4) at the dose determined from the data from Cohort 1 and 2. GSK2256294 capsules will be available in 1, 5, 25 mg dose strength.
Drug: Placebo — Matching placebo will be administered once daily (cohorts 1 and 2); and once or twice daily (cohorts 3 and 4).

SUMMARY:
This study is the First Time in Human Study for GSK2256294 and will evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of single and repeat oral doses of GSK2256294 administered to healthy male volunteers (Cohort 1) and otherwise healthy adult male moderately obese smokers (Cohorts 2 to 4). Cohorts 1 and 2 will enrol 12 subjects each and each subject will take part in four study periods. All subjects will receive placebo regimen and three dosing regimens of GSK2256294 in a specified sequence (planned doses 2 mg, 6 mg and 18 mg in Cohort 1 and 15 mg, 40 mg and 100 mg in Cohort 2). Each study period will be followed by a Wash-out period of 7 to 14 days in Cohort 1 and up to 4 weeks in Cohort 2. During each study period subjects will be in-house from Day -1 until the 48 hours post dose assessments have been completed. Subjects will return to the unit as out-patients for remaining post-dose assessments. Subjects will then be followed for 7 to 14 days in Cohort 1 and up to 3 to 4 weeks in Cohort 2. Total duration of the study for Cohort 1 will be 98 days and for Cohort 2 it will be up to 144 days. Cohort 3 and 4 will each recruit 15 subjects. For Cohorts 3 and 4, each subject will take part in one treatment period of 18 days (Day-1 to Day 17) with dosing from Day 1 to Day 14. Subjects will then be followed for 7 to 14 days. Total duration of the study for Cohort 3 and Cohort 4 will be 67 days. Dose selection for Cohorts 3 and 4 will be based on the safety, PK profile and enzyme inhibition obtained in Cohorts 1 and 2. This study will also evaluate the evidence for a functional effect of soluble Epoxide Hydrolase (sEH) in a forearm blood flow (FBF) model.

ELIGIBILITY:
Inclusion Criteria:

* Suitable for cannulation and with adequate venous access.
* 12 lead ECG without any clinically significant abnormality as judged by the Investigator, and ECGs QTcF (QT interval was corrected using Fridericia's formula)<=450 milliseconds (msec) determined by the average of triplicate ECGs.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter outside the reference range for the population being studied may be included only if the Investigator agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Consultation with the medical monitor is required.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Male between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Male subjects must agree to use one of the approved contraception methods This criterion must be followed from the time of the first dose of study medication until the follow-up visit.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* For Cohort 1 Only: Subjects should have blood pressure (BP) <=130/80; body weight >=60 kilograms (kg) and body mass index (BMI) within the range 19 to 25 kilogram/meter squared (kg/m^2) (inclusive); subjects should be non-smokers, which for this study is defined as having smoked <100 cigarettes or <1 pack per year in their lifetime.
* For Cohorts 2 to 4 Only: Subjects must have smoked in the 12 month period preceding the screening visit. Smoking is defined as >=10 cigarettes/day for at least the preceding 1 year, and have a >5-pack year history. [number of pack years = (number of cigarettes per day/20) x number of years smoked]; having body weight >=60 kg and BMI within the range 28 to 35 kg/m^2 (inclusive); and BP <=140/90.
* Cohorts 3 and 4 Only: Palpable brachial artery in the non-dominant and/or dominant hands, as assessed by a clinician at screening.

Exclusion Criteria:

* Subjects with any history of a carcinoma.
* Participants who have had previous vasovagal events secondary to any painful stimulus e.g. venepuncture or have a phobia of blood.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Significant cardiac, pulmonary, metabolic, renal, gastrointestinal or other conditions that in the opinion of the investigator and/or GlaxoSmithKline (GSK) medical monitor, places the subject at an unacceptable risk as participant in this trial. Patients with asthma or diabetes are excluded.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody at screening.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males. One unit is equivalent to 8 g of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* The use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator or GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety. Other concomitant medication may be considered on a case by case basis by the GSK Medical Monitor.
* History of sensitivity to any of the study medications and challenge agents, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* For Cohorts 2 to 4 Only: Smokers who require a cigarette within 30 minutes after they wake in the morning, or cannot abstain from smoking for approximately 5 hours; or subjects with symptomatic asthma requiring regular inhaled or oral steroids and bronchodilators.; or subjects who are currently on statins or have been on statins within 3 months prior to the first dose of study medication.
* For Cohorts 3 and 4 Only: Subjects who are unable to lie still for the duration of the forearm study (up to 3 hours).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2013-01-16 (Actual); Primary Completion 2014-05-01 (Actual); Study Completion 2014-05-01 (Actual)

PRIMARY OUTCOMES:
Safety of single oral doses of GSK2256294 assessed by clinical monitoring of vital signs (Cohort 1). | Up to 98 days.
  Vital signs include systolic blood pressure, diastolic blood pressure, and pulse rate. Vital signs will be collected with the subject semi-supine and after they have been resting for 5 minutes.
Safety of single oral doses of GSK2256294 assessed by clinical monitoring of vital signs (Cohort 2). | Up to 144 days.
  Vital signs include systolic blood pressure, diastolic blood pressure, and pulse rate. Vital signs will be collected with the subject semi-supine and after they have been resting for 5 minutes.
Safety of single oral doses of GSK2256294 assessed by clinical monitoring of Electrocardiogram (Cohort 1). | Up to 98 days.
  12-lead electrocardiograms (ECGs) will be obtained at each time point during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTcF intervals. ECGs will be obtained in the semi-supine position after the subject has been resting for at least 5 minutes.
Safety of single oral doses of GSK2256294 assessed by clinical monitoring of Electrocardiogram (Cohort 2). | Up to 144 days.
  12-lead electrocardiograms (ECGs) will be obtained at each time point during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTcF intervals. ECGs will be obtained in the semi-supine position after the subject has been resting for at least 5 minutes.
Safety of repeat oral doses of GSK2256294 assessed by clinical monitoring of vital signs (Cohort 3 and 4). | Up to 67 days
  Vital signs include systolic blood pressure, diastolic blood pressure, and pulse rate. Vital signs will be collected with the subject semi-supine and after they have been resting for 5 minutes.
Safety of repeat oral doses of GSK2256294 assessed by clinical monitoring ECG (Cohort 3 and 4). | Up to 67 days.
  12-lead ECGs will be obtained at each time point during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTcF intervals. ECGs will be obtained in the semi-supine position after the subject has been resting for at least 5 minutes.
Safety of single oral doses of GSK2256294 assessed by clinical laboratory assessments (Cohort 1 ). | Up to 98 days.
  Safety data will include assessments of clinical laboratory tests (hematology, clinical chemistry and urinalysis).
Safety of single oral doses of GSK2256294 assessed by clinical laboratory assessments (Cohort 2). | Up to 144 days.
  Safety data will include assessments of clinical laboratory tests (hematology, clinical chemistry and urinalysis).
Safety of repeat oral doses of GSK2256294 assessed by clinical laboratory assessments (Cohort 3 and 4). | Up to 67 days.
  Safety data will include assessments of clinical laboratory tests (hematology, clinical chemistry and urinalysis).
Safety of single oral doses of GSK2256294 assessed by number of participants with adverse events (Cohort 1). | Up to 98 days.
  Adverse events (AEs) will be recorded from the start of Study Treatment until the follow-up contact.
Safety of single oral doses of GSK2256294 assessed by number of participants with adverse events (Cohort 2). | Up to 144 days.
  AEs will be recorded from the start of Study Treatment until the follow-up contact.
Safety of repeat oral doses of GSK2256294 assessed by number of participants with adverse events (Cohort 3 and 4). | Up to 67 days.
  AEs will be recorded from the start of Study Treatment until the follow-up contact.

SECONDARY OUTCOMES:
Composite of PK parameters following single dose of GSK2256294. | PK samples will be collected at pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72 hours post dose in each treatment period.
  PK parameters include: maximum observed plasma concentration (Cmax), time to Cmax (tmax), area under the plasma concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration (AUC [0-t]) and from time zero extrapolated to infinite time (AUC[0-infinity]), apparent terminal phase half-life (t1/2). AUC (0-infinity) or area under the concentration-time curve over the dosing interval (AUC[0-tau]) and Cmax following single and repeat doses may be used for assessment of dose proportionality.
Composite of PK parameters following repeat doses of GSK2256294. | Up to Day 17 in Cohort 3 and 4
  PK parameters include: Cmax, tmax, (AUC [0-t]), (AUC [0-infinity]), (t1/2). AUC (0-infinity) or (AUC [0-tau]) and Cmax following single and repeat doses may be used for assessment of dose proportionality. Trough concentration (Ctau) samples collected on the specified days may be used to assess attainment of steady state.
Percent inhibition of sEH enzyme activity in whole blood after single oral dose of GSK2256294 as a measure of PD effect. | Plasma samples will be collected at pre-dose, 1, 2, 6, 8, 12, 24, 48, and 72 hours post dose in Cohort 1 and 2.
  Percent inhibition of soluble sEH enzyme activity in whole blood will be measured from plasma samples. GSK2256294 is a potent and reversible inhibitor of sEH and this will be evaluated to determine the PD effect of GSK2256294 on sEH enzyme activity.
Percent inhibition of sEH enzyme activity and Leukotoxin : leukotoxin-diol ratio in plasma after repeat oral doses of GSK2256294 . | Up to Day 17 in Cohort 3 and 4
  The PD inhibitory effect of repeat oral doses of GSK2256294 on sEH inhibition in the study population will be investigated via the sEH enzyme inhibition assay and the ratio of leukotoxin to leukotoxin diol data subject to data available from the study. Samples will be collected to measure sEH enzyme inhibition and the ratio of substrate to product for biomarkers: leukotoxin: leukotoxin diol ratio
Exposure-response relationship between the blood concentration of GSK2256294 and sEH enzyme inhibition, leukotoxin : leukotoxin-diol ratio (if data permit) following single dose of GSK2256294. | Plasma samples will be collected at pre-dose, 1, 2, 6, 8, 12, 24, 48, and 72 hours post dose in cohort 1 and 2.
  Based on the availability of data, a PK/PD model will be attempted to explain the dose response (exposure response) relationship between GSK2256294 and the various biomarkers analyzed in the study.
Exposure-response relationship between the blood concentration of GSK2256294 and sEH enzyme inhibition, leukotoxin : leukotoxin-diol ratio (if data permit) following repeat doses of GSK2256294. | Up to Day 17 in cohort 3 and 4.
  Based on the availability of data, a PK/PD model will be attempted to explain the dose response (exposure response) relationship between GSK2256294 and the various biomarkers analyzed in the study.
Change from baseline forearm blood flow relative to the preceding challenge agent, as measured by venous occlusion plethysmography. | Baseline (screening) and Day 1 and Day 14 in Cohort 3 and 4.
  A plethysmograph is an instrument for measuring changes in volume within an organ or whole body (usually resulting from fluctuations in the amount of blood or air it contains). It will be used to determine the effects of GSK2256294 and placebo on endothelium-dependent and independent vasodilatation.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Yang L, Cheriyan J, Gutterman DD, Mayer RJ, Ament Z, Griffin JL, Lazaar AL, Newby DE, Tal-Singer R, Wilkinson IB. Mechanisms of Vascular Dysfunction in COPD and Effects of a Novel Soluble Epoxide Hydrolase Inhibitor in Smokers. Chest. 2017 Mar;151(3):555-563. doi: 10.1016/j.chest.2016.10.058. Epub 2016 Nov 21. PMID 27884766
- [Derived] Lazaar AL, Yang L, Boardley RL, Goyal NS, Robertson J, Baldwin SJ, Newby DE, Wilkinson IB, Tal-Singer R, Mayer RJ, Cheriyan J. Pharmacokinetics, pharmacodynamics and adverse event profile of GSK2256294, a novel soluble epoxide hydrolase inhibitor. Br J Clin Pharmacol. 2016 May;81(5):971-9. doi: 10.1111/bcp.12855. Epub 2016 Jan 17. PMID 26620151
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 114068 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/114068?search=study&search_terms=114068#rs
- Available data/document: Study Protocol: 114068 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114068 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114068 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114068 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114068 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114068 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114068 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register